CLINICAL TRIAL: NCT06639737
Title: Effect of Preoperative Stroke Volume Optimization Using Transthoracic Echocardiography on Arterial Hypotension Following Induction of Intravenous Anesthesia. A Prospective, Double Blinded Randomized Study.
Brief Title: Preoperative Blood Volume Optimization Using Transthoracic Echocardiography
Acronym: EchOptimal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID-RCB 2024-A01292-45
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia; Anesthesia Complication; Anesthesia Induction; Arterial Hypotension
Keywords: preoperative stroke volume optimization echocardiography; arterial hypotension; general anesthesia; transoesophageal doppler; sub aortic velocity time integral
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): Standard care : total intravenous anesthesia followed by stroke volume optimization using oesophageal doppler
  Interventions: Procedure: Post induction stroke volume optimization
- preoperative echography (Experimental): Stroke volume optimization using transthoracic echocardigraphy (sub aortic velocity time integral) before induction of total intravenous anesthesia
  Interventions: Procedure: preoperative stroke volume optimization

INTERVENTIONS:
Procedure: preoperative stroke volume optimization — Stroke volume optimization using transthoracic echocardigraphy (sub aortic velocity time integral) before induction of total intravenous anesthesia. Fluids bolus of 250 ml of cristalloids will be successively administered until the sub aortic velocity time integral increase will be < 10%
  Arms: preoperative echography
Procedure: Post induction stroke volume optimization — Optimization of stroke volume following induction of general anesthesia using oesophageal stroke volume measurement. 250 ml bolus of cristalloids succesively administered until the stroke volume increase <10%
  Arms: control

SUMMARY:
Immediately following the induction of general anesthesia, arterial hypotension may occur with an incidence of about 40% in patients classified as ASA 3 or 4. Perioperative arterial hypotension is associated with increased perioperative morbidity and mortality. The increased mortality associated with perioperative arterial hypotension has been reported up to 30 and 90 days after surgery. This association appears to be both dose-dependent and time-dependent (severity and duration of arterial hypotension).

EchOptimal study aims to determine whether non invasive preoperative stroke volume optimization using transthoracic echocardiography (TTE) can reduce the incidence and severity arterial hypotension following induction of general anesthesia.

This is prospective, randomized, controlled, double blinded study approved by ethics comittee.

The primary objective of this study is to compare the incidence of arterial hypotension (mean arterial pressure < 65 mmHg) within the first 15 minutes following the induction of general anesthesia, between 2 groups :

* standard current care (stroke volume optimized after induction of general anesthesia using oesophageal doppler) and
* preopertaive stroke volume optimization using transthoracic echocardiography measument of subaortic velocity time integral.

DETAILED DESCRIPTION:
The pre-inclusion visit consists of a preoperative evaluation of the patient in the emergency operating room. This evaluation is conducted by an anesthesiologist for all patients requiring surgical care in the emergency operating room.

This evaluation is structured similarly to a pre-anesthetic consultation conducted by an anesthesiologist for scheduled surgery. During this preoperative evaluation, the patient's medical and surgical history, current treatments, and possible allergies are collected. A targeted clinical examination is also performed.

After this evaluation, the anesthesiologist analyzes the risks posed by the patient and the specific risks associated with surgery and anesthesia to define the best perioperative strategy.

Surgical interventions are classified into three categories of postoperative cardiovascular risk (low, intermediate, or high) for cardiovascular complications within 30 days post-surgery, according to the table provided by French and European recommendations.

During this consultation, patients eligible for the study (ASA classification 3 or 4, requiring general anesthesia for intermediate or high-risk surgery) will be identified.

After verifying the inclusion/exclusion criteria, the patient will be informed about the study, its course, objectives, and constraints.

An information letter will be given to the patient, and their informed consent will be collected in writing.

The pre-inclusion and inclusion visits will thus take place at the same time.

2. Inclusion visit (V0):

This visit is conducted alongside the pre-inclusion visit:

* Verification of inclusion/non-inclusion criteria by the investigator.
* Patient information regarding the study, its procedures, constraints, and foreseeable risks.
* Presentation of the information letter and obtaining of written informed consent after ensuring the patient's full understanding of the proposed protocol and answering all questions.
* Collection of main medical history and concurrent treatments.
* Clinical examination with vital signs.
* Explanation of the study procedures.

  3. Practical implementation of the protocol - patient management:

After inclusion (as per paragraphs 1 and 2 above), all patients will undergo standard perioperative monitoring:

* 5-lead electrocardiogram (IntelliVue MP 70, Philips HealthCare, Amsterdam, Netherlands).
* Pulse oximetry.
* Direct and continuous blood pressure measurement using a catheter inserted under local anesthesia into the radial artery (right or left), after verifying no contraindications. The catheter will be connected to a pressure transducer calibrated at the fifth intercostal space at the mid-axillary line.
* Bispectral index (BIS™ Quatro Sensor, Covidien, Dublin, Ireland) to monitor anesthesia depth, keeping values within the recommended range (between 45 and 55).
* Accelerometer (Philips IntelliVue NMT, Philips HealthCare, Amsterdam, Netherlands) placed on the thumb opposite the continuous blood pressure measurement site to monitor the effects of neuromuscular blocking agents (curare).

Before entering the operating room (in the recovery room of the emergency operating block), the patients will undergo the following:

* Control group : A transthoracic echocardiography (TTE) without volume optimization, performed as recommended for preoperative evaluation of ventricular and valvular function. This TTE will be carried out by an experienced operator independent of the patient's care.
* Experimental group : A TTE with volume optimization as explained earlier, performed by an experienced operator independent of the patient's care.

For all patients, the independent operator performing the TTE will share the collected data (ventricular and valvular function) with the anesthesiologist in charge of the patient. This data, which is important for patients with the included profile, will be collected as recommended and documented in a standardized report in the anesthesia consultation software.

In the operating room, the patient management will follow best practices for anesthesia and intensive care based on the patient profile, including:

* Comfortable patient positioning and warming using a forced-air warming blanket (BairHugger™, 3M France, Cergy-Pontoise, France).
* Pre-oxygenation with a target expired O2 fraction above 90% before induction of general anesthesia.
* Induction of general anesthesia via intravenous injection using automated syringes with target-controlled anesthesia software with propofol and remifentanil. The depth of anesthesia will be adjusted according to the bispectral index values.
* Administration of curare.
* Orotracheal intubation and mechanical ventilation following perioperative protective ventilation recommendations adapted to the patient (FiO2 40%, tidal volume 6-8 mL/kg of ideal body weight, PEEP

  * 5 to +8 cmH2O).
* Insertion of the esophageal Doppler probe (Cardio-Q, Gamida, Eaubonne, France) and urinary catheter.
* Volume optimization for both groups following current recommendations, using stroke volume measurements from the esophageal Doppler and simultaneous measurement of the subaortic time-velocity integral (ITVSAo) with TTE.

Throughout the induction of anesthesia and during the 15 minutes corresponding to the collection of the primary outcome, an independent investigator not involved in patient care will record all the necessary data.

4. Follow-up evaluations during the study (V1, V2, etc.): No additional blood samples are required for this study. A preoperative TTE called a "preoperative screening" (FOCUS exam) is proposed preoperatively for patients meeting the inclusion criteria of this study to evaluate their overall cardiac function before the intervention [15] (Class IIB, Level of Evidence B recommendation from the 2022 European Society of Cardiology guidelines on the assessment and management of patients undergoing non-cardiac surgery). As a result, the proportion of TTEs performed "in addition" compared to standard care will be minimal or none and can only be beneficial for preoperative assessment.

However, volume optimization is not routinely performed before the induction of general anesthesia as described earlier (in the summary and context paragraphs). This optimization does not require blood samples but involves a guided administration of crystalloids (currently, this administration is often empirical and not measured).

The echocardiography machines used will be those already present in the operating room (no additional equipment is required for this study).

5. End-of-study evaluation: The follow-up ends 15 minutes after the completion of general anesthesia induction.

An analysis of all data between the start of induction and 15 minutes after the end of induction will be performed.

6. Long-term follow-up evaluation: No long-term follow-up evaluation.

10. Data to be collected

All data recorded by the monitoring devices of a patient during general anesthesia will be noted. This includes:

Before the induction of general anesthesia:

* Data from the preoperative evaluation of the patient (age, weight, height, chronic conditions, chronic treatments, ASA classification, operative indication, systolic, diastolic, and mean blood pressure, heart rate, peripheral oxygen saturation).
* TTE data including the subaortic time-velocity integral (ITVSAo).
* Data on the volume optimization performed in the experimental group (volume of crystalloids administered, type of crystalloid, repeated measurements of ITVSAo, blood pressure, heart rate, peripheral oxygen saturation).
* Time required for volume optimization (from the placement of the echocardiography probe to the end of the last administration of crystalloids).

During the induction of general anesthesia and for the 15 minutes following the initiation of controlled ventilation:

* Maximum cerebral targets for propofol and remifentanil used with the target-controlled intravenous anesthesia syringe.
* The highest and lowest systolic, diastolic, and mean blood pressure.
* Duration during which a blood pressure < 65 mmHg is measured (since the blood pressure is measured continuously, this duration is assessed in 1-minute intervals).
* The highest and lowest respiratory variation in pulse pressure.
* The highest and lowest heart rate.
* The highest and lowest oxygen saturation.
* The highest and lowest expired CO2 levels.
* The highest, lowest, and average bispectral index over 15 minutes.
* Data from the volume optimization after the induction of general anesthesia obtained via esophageal Doppler (stroke volume, corrected ejection time, peak velocity), repeated measurements of blood pressure, heart rate, and peripheral oxygen saturation.
* Volume of crystalloids administered for volume optimization after induction.
* Vasopressor medications administered (name and total doses).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older,
* Affiliated with social security,
* Informed about the study and having signed the informed consent form,
* Requires surgical intervention under general anesthesia,
* Intermediate or high risk of cardiovascular events within 30 days,
* ASA phyiscal status Classification 3 or 4

Exclusion Criteria:

- Pregnant or breastfeeding women,

* Patients under guardianship, curatorship, judicial protection, or legal protection,
* Minors,
* Patients with contraindications to intravenous induction with Propofol and Remifentanil,
* Patients not fasting at the time of surgery,
* Patients with an immediate life-threatening emergency or requiring surgery without delay to ensure survival,
* Patients with contraindications for placing an arterial pressure catheter in the radial artery: bilateral negative Allen's test indicating absence of ulnar collateral circulation, Raynaud's syndrome, Buerger's disease, severe dyslipidemias,
* Patients with characteristics making the measurement of ITVSAo uninterpretable: atrial fibrillation, non-sinus electrocardiogram, severe valvulopathy, documented right or left heart failure,
* Patients under general anesthesia before arrival in the operating room,
* Patients receiving aminergic support before anesthetic induction,
* Patients requiring rapid sequence induction,
* Patients treated with ACE inhibitors/ARBs who have not discontinued the treatment on the day of the procedure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
arterial hypotension | From enrollment to 15 min after orotracheal intubation during total intravenous anesthesia
  Incidence (%) of arterial hypotension (mean arterial pressure < 65 mmHg) within 15 minutes following induction of general anesthesia.
  Blood pressure will be continuously measured using a radial arterial pressure catheter placed before induction of anesthesia in all patients.

SECONDARY OUTCOMES:
technical failure of preoperative stroke volume optimization | From enrollment to 15 min after orotracheal intubation during total intravenous anesthesia
  Proportion (%) of patients in whom volume preoperative stroke volume optimization could not be performed.
duration of arterial hypotension | From enrollment to 15 min after orotracheal intubation during total intravenous anesthesia
  Cumulative duration (in minutes) of arterial hypotension from the start of anesthetic drug administration until 15 minutes after orotracheal intubation
lowest mean arterial hypotension | From enrollment to 15 min after orotracheal intubation during total intravenous anesthesia
  Lowest mean arterial pressure (in mmHg)measured.
vasoactive drugs administration | From enrollment to 15 min after orotracheal intubation during total intravenous anesthesia
  Proportion (%) of patients requiring vasopressor during the measurement period.
cristalloids volume | From enrollment to 15 min after orotracheal intubation during total intravenous anesthesia
  Total volume of cristalloids require during the measurment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Universty Hospital of Caen, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided